CLINICAL TRIAL: NCT03577353
Title: Dual-task Training Using Virtual Reality: Influence on Walking and Balance in Post Stroke Survivors
Brief Title: Dual-task Training Using Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loewenstein Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0001-13-LOE
Record Dates: First submitted 2018-05-21; First posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental-DTW (Experimental): The intervention of the experimental group was based on dual-task treadmill walking while using the Virtual Reality (VR) tool.
  Interventions: Behavioral: Dual Task Walking (DTW)
- Control- TMW (Active Comparator): The intervention of the control group was based on single-task treadmill walking.
  Interventions: Behavioral: Single-task Treadmill Walking (TMW)

INTERVENTIONS:
Behavioral: Dual Task Walking (DTW) — Each training session began with 8 min of general warm-up and 2 min walk around the gym. Then, for safety reasons, the participants were attached to a harness. The participants began walking slowly on the treadmill for 3 min. In the following phases the participants walked at the same speed, while training with 3 VR games. Each session lasted 3 min, and 3 min of single walking was performed between VR sessions. After the final VR session, 2 min of single-task walking was performed in order to allow for recovery. The time walked in each trial from the starting point to the destination was kept constant at 20 min.
  Arms: experimental-DTW
Behavioral: Single-task Treadmill Walking (TMW) — this intervention, participants performed 8 min of general warm-up and 2 min walk around the gym, and then continued to walk for another 20 min on the treadmill at a speed that was equivalent to the intensity of 60%-70% of their heart rate reserve.
  Arms: Control- TMW

SUMMARY:
The purpose of the study was to investigate the feasibility of using a virtual reality- based dual task training of upper extremity tracking while treadmill-walking, to improve walking and balance performance in post stroke survivors

ELIGIBILITY:
Inclusion Criteria:

* With hemiplegia after a stroke for at least a year since the incident.
* Range age 40-80.
* Without medication or with stabilized medication.
* Use ankle-foot orthosis or no splint at all.

Exclusion Criteria:

* Severe cardiac problems
* A score less than 25 in the Mini-Mental test.
* Fractures or severe orthopedic limitations that do not allow for training, and which have occurred over the last six months.
* More than three falls in the past year before participating in the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-10-30 (Actual); Primary Completion 2016-08-18 (Actual); Study Completion 2017-11-26 (Actual)

PRIMARY OUTCOMES:
change in 10-meter walking test across pre, post and follow-up time points. | Pre-intervention time: one week before the intervention period (4 week).Post intervention time:immediately after the intervention. Follow-up time: 4 weeks after intervention
Change in Timed up and go across pre, post and follow-up time points. | Pre-intervention time: one week before the intervention period (4 week).Post intervention time:immediately after the intervention. Follow-up time: 4 weeks after intervention
Change in Functional Reach Test across pre, post and follow-up time points. | Pre-intervention time: one week before the intervention period (4 week).Post intervention time:immediately after the intervention. Follow-up time: 4 weeks after intervention
Change in Activities-specific Balance Confidence (ABC) Scale | Pre-intervention time: one week before the intervention period (4 week).Post intervention time:immediately after the intervention. Follow-up time: 4 weeks after intervention
  Activities-specific Balance Confidence (ABC) Scale is a 16-item questionnaire/survey. Each item is rated from 0% (no confidence) to 100% (complete confidence). Elderly respondents are asked to rate their confidence that they will lose their balance or become unsteady in the course of daily activities. ABC is an 11-point scale and ratings should consist of whole numbers (0-100) for each item. Participants should indicate their level of confidence in doing an activity without losing balance or becoming unsteady by choosing one of the percentage points on the scale from 0%-100%. Total the ratings (possible range = 0 to 1600) and divide by 16 to get each subject's ABC score. Scores lower than 50 indicate a low level of functioning, scores above 50 but below 80 indicate a medium level, and those over 80 indicate a high level of functioning.
Change in The Berg Balance Scale (BBS) across pre, post and follow-up time points. | Pre-intervention time: one week before the intervention period (4 week).Post intervention time:immediately after the intervention. Follow-up time: 4 weeks after intervention
  14-item scale designed to measure balance of the older adult in a clinical setting. A five-point ordinal scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function.Total Score = 56. 41-56 = low fall risk, 21-40 = medium fall risk, 0 -20 = high fall risk.

CONTACTS AND LOCATIONS:
Overall Officials: Yeshayahu Hutzler, Ph.D., Study Director — Graduate School Academic College at Wingate
Locations (1):
- The Academic College at Wingate, Netanya, Israel

IPD SHARING:
Plan to Share IPD: Undecided